CLINICAL TRIAL: NCT05113602
Title: Validation of the EEG Signal Quality Measured by the URGOnight Device and Comparison With a Clinical Device
Acronym: SIGMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Urgotech (Industry)
Collaborators: ESPCI Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SIGMA
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volonteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simultaneous acquisition of EEG signals (Experimental)
  Interventions: Device: URGOnight; Device: Enobio

INTERVENTIONS:
Device: URGOnight — EEG dry electrodes portable device
Device: Enobio — EEG wet electrodes portable device

SUMMARY:
The electroencephalogram or EEG is a painless and non-invasive exploratory examination routinely performed in clinical and experimental medicine and has various applications. It is therefore relevant to develop application-specific EEG measurement devices.

The clinical development of therapies based on brain control has led to the emergence of numerous EEG devices that aim to allow mobile, autonomous, and easy use for users.

Data from the literature have proven the ability of neurofeedback (a form of biofeedback in which subjects respond to a display of their own brainwaves in order to improve their health or performance) to improve brain function in healthy or pathological subjects.

These therapeutic applications are offered in hospital settings with conventional systems and in the presence of a therapist.

The EEG measurement device URGOnight was developed with the aim of offering autonomous neurofeedback exercises at home. URGOnight is a portable device. It uses passive electrodes (which do not send an electric current) and so-called dry electrodes, i.e. no gel or conductive paste is required.

Therefore, the SIGMA study aims to evaluate the quality of the EEG signal collected by URGOnight and compare it with an electroencephalography device commonly used in clinical and research settings.

We will also evaluate the quality of the brain wave measurement usually retained in comparative studies of EEG systems.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Head circumference between 52 and 62 centimeters
* Affiliated or beneficiary of a social security system
* Protected persons in the sense of article L.1121-9 of the Public Health Code.

Exclusion Criteria:

* According to declarative :
* Use of medication or drugs with a possible effect on cognitive performance, such as benzodiazepines, antidepressants and antipsychotics
* Epilepsy
* The experimenter cannot get a good signal between the scalp and the electrodes at the beginning of the experiment (for example because of the type of hair or for any other technical reason).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
effectiveness of the URGOnight device in detecting brain signals triggered by eye closure in the Alpha band (8-12 Hz) in comparison with the Enobio 20 device. | 5 min recording

SECONDARY OUTCOMES:
To compare the measurement performed by URGOnight to the measurement performed by the Enobio 20 device of Visual evoked potentials SSVEP at 4, 8, 10, 13, 15 and 20 hertz | 5 min recording
To compare the measurement performed by URGOnight to the measurement performed by the Enobio 20 device of SMR rhythm | 10 min recording
To compare the measurement performed by URGOnight to the measurement performed by the Enobio 20 device of Individual Alpha frequencies | 10 min recording

OTHER OUTCOMES:
Optimize protocols to identify and distinguish individual Alpha and SMR peaks | 20 min recording

CONTACTS AND LOCATIONS:
Locations (1):
- ESPCI, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided